CLINICAL TRIAL: NCT01150968
Title: An Educational Intervention to Improve Resident Comfort With Communication at the End of Life
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, San Francisco (Other)
Responsible Party: Bernard Lo, MD, UCSF
Allocation: Not Applicable | Model: Single Group | Masking: None
Other Study IDs: 10035736
Record Dates: First submitted 2010-06-24; First posted 2010-06-25 (Estimated); Last update posted 2011-02-10 (Estimated); Status verified 2011-02

CONDITIONS: End of Life Communication

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Internal Medicine Residents (Experimental): All UCSf Internal Medicine residents for 2009-2010
  Interventions: Behavioral: End of life education

INTERVENTIONS:
Behavioral: End of life education — Residents will participate in one hour, case-based, interactive teaching sessions on end of life communication.

SUMMARY:
The purpose of this study is to investigate whether the addition of teaching on communication at the end of life to the pre-existing resident curriculum will positively impact residents' knowledge and attitudes regarding communication at the end of life.

DETAILED DESCRIPTION:
Previous research has demonstrated a lack of resident training in communication at the end of life. This can lead to anxiety on the part of residents and poor experiences with these conversations. Residents at UCSF, and affiliated sites, participate in a daily formal teaching session from 12-1 pm and an informal case conference, known as Morning Report, from 7:30-8:30 am (8-9 am at VAMC). We propose to administer a pre-intervention survey to residents to assess knowledge and attitudes regarding communication at the end of life. Over two months, residents will receive one lecture during the noon session. Clinical cases will be presented for discussion during three sessions of morning report. All sessions are voluntary and take place at all three training sites, UCSF, SFGH, and the VAMC. As residents rotate every two months between the inpatient and outpatient settings, the intervention will be repeated once to ensure that the majority of residents have the opportunity to participate. A post-intervention survey, identical to the pre-intervention survey, will be administered to assess for impact of the educational intervention. This project only involves UCSF Internal Medicine residents. No patients will be involved in this study.

ELIGIBILITY:
Inclusion Criteria:

* UCSF internal medicine resident

Exclusion Criteria:

* Not UCSF internal medicine resident

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 166 (Estimated)
Dates: Start 2010-03; Primary Completion 2010-06 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Self-efficacy | 90 days
  Residents participating in the intervention will demonstrate increased self-efficacy for end of life conversations.

CONTACTS AND LOCATIONS:
Locations (1):
- UCSF Program in Medical Ethics, San Francisco, California, United States